CLINICAL TRIAL: NCT00862537
Title: An Open-label Extension Study for Subjects Previously Treated Either in Pilot I or Pilot II Studies of the Application of Magnetic Fields Using the Resonator for the Treatment of Parkinson's Disease.
Brief Title: Evaluation of Long-term Effect of Resonator Therapy on Parkinson's Disease (PD)
Status: Completed | Type: Observational
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: pico-tesla Magnetic Therapies, LLC, pico-tesla Magnetic Therapies, LLC
Other Study IDs: PD Ext
Record Dates: First submitted 2008-10-22; First posted 2009-03-17 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Active Resonator magnetic field therapy: Administration of active magnetic fields with the Resonator Device
  Interventions: Device: Resonator Device

INTERVENTIONS:
Device: Resonator Device — active pico-tesla magnetic fields treatment for Parkinson's disease individuals

SUMMARY:
An extension study for subjects with prior participation in previous resonator studies using low level magnetic fields to treat some of the symptoms of idiopathic Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in pico-tesla pilot studies: NCT00779155 & NCT00863226
* Willing and able to abstain from partaking in non-essential new treatments for Parkinson's disease symptoms during the course of participation of the study.
* Will and able to abstain from all non-essential new medications that could affect PD and/or any of its associated symptoms for the duration of the study.
* Willing to notify the investigator right away of any changes in medication use or therapies that is prescribed and deemed necessary by the subjects physicians.
* Adequate contraceptive measures for female subjects
* Capable of giving full written informed consent

Exclusion Criteria:

* Not a participant in IRC#'s 07102 or 07021
* No active brain tumors, strokes, hydrocephalus
* Chronic pain not associated with PD
* Any other condition which might prevent subject from comfortably sitting for 1.5 hours
* Consumption of medications that can produce Parkinsonism type symptoms
* Major psychiatric disturbance
* Epilepsy
* HIv and other autoimmune disorders
* Cancer within last 2 years
* History of ECt
* Diabetic neuropathy
* Uncontrolled HTN
* Advanced Pulmonary disease
* Known heart conditions such as repetitive history of cardiac arrythmias
* Previous surgeries for PD
* Prosthetics comprised of ferrous materials
* Stents, only where there is also cardiac arrythmias, CHF, advanced valvular stenosis, unstable vital signs, extensive ischemic damage to heart muscle as a result of one or more heart attacks.
* Pacemakers
* Uncontrolled, unstable, or untreated medical illnesses which might potentially significantly affect the patient's health in the opinion of the investigator
* Consumption of more than 21 alcoholic drinks per week
* Pregnant, breast feeding or planning pregnancy
* Developmental disability or cognitive impairment
* Inability to maintain regular medication regime
* Inability to abstain from partaking in new non-essential PD tx., or medications
* Not willing to report physician mandated changes in medication and/or treatment

Ages: 30 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previous participants enrolled in one of two prior pico-tesla Magnetic Therapies Resonator device studies using magnetic fields for treating Parkinson's Disease (PD) symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry I Jacobson, PhD., DMD., Principal Investigator — pico-tesla Magnetic Therapies, LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Resontaor Device Therapy: active pico-tesla magnetic fields Resonator device therapy
Period: Overall Study
Arm/Group | Active Resontaor Device Therapy
Started | 18
Completed | 11
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Active Resontaor Device Therapy
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Parkinson's Disease Questionnaire-39 Single Index Score (PDQ-39SI)From Baseline to Study Endpoint of 11 Months
Description: The Parkinson's Disease Questionnaire (PDQ-39) is a 39-item quality of life questionnaire for patients with Parkinson's Disease (PD) that evaluates the 8 dimensions of mobility, activities of daily living, emotional well-being, stigma, social support, cognition, and communication. The PDQ-39 Single Index (SI) score is the weighted addition of scores on all 8 dimension and ranges from 0 (no disease impact) to 100 (severe disease impact).
Time Frame: baseline and 11 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Resontaor Device Therapy
Number analyzed (Participants) | 18
scores on a scale | 4.96 (1.1)

ADVERSE EVENTS:
Arm/Group | Active Resontaor Device Therapy
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes